CLINICAL TRIAL: NCT06766448
Title: Robotic Training in the Management of Adhesive Capsulitis: a Randomized Controlled Trial
Brief Title: Effectiveness of Instrumental Rehabilitation in Patients With Adhesive Capsulitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mohammed V Souissi University (Other)
Responsible Party: Principal Investigator, SARA SKALLI, assistant professor, Mohammed V Souissi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C63-20
Record Dates: First submitted 2025-01-04; First posted 2025-01-09 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Adhesive Capsulitis of the Shoulder
Keywords: adhesive capsulitis; rehabilitation; robotic training
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention group (Experimental): the intervention group will receive robotic training
  Interventions: Other: robotic training
- control group (Active Comparator): control group will receive conventionnal rehabilitation
  Interventions: Other: conventionnal rehabilitation

INTERVENTIONS:
Other: robotic training — continuous passive mobilization and robotic therapy on armeo sping
  Arms: intervention group
Other: conventionnal rehabilitation — rehabilitation sessions with a physiotherapist
  Arms: control group

SUMMARY:
The aim of this study is to evaluate the effectiveness of robotic training compared to conventional rehabilitation in patients with AC.

DETAILED DESCRIPTION:
Nowadays, rehabilitation focuses on functional work during physiotherapy sessions to improve the patient's autonomy.

In the era of new technologies, robotics and virtual reality have shown great interest in functional rehabilitation and cortical reorganization.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years of age
* Shoulder pain and/or movement limitation
* Idiopathic AC or associated with confirmed systemic disease (e.g., diabetes or dyslipidemia)

Exclusion Criteria:

* Cognitive impairment
* History of surgery
* Fracture or dislocation of the shoulder
* History of shoulder tendinopathy
* History of inflammatory or degenerative disease
* Infection
* Neurological disease (Parkinson's disease, stroke, multiple sclerosis, neurological
* Manipulation under anesthesia, hydro dilation, platelet rich plasma or hyaluronic acid infiltration within the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-03-23 (Actual); Primary Completion 2025-01-02 (Actual); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
shoulder fonction using Shoulder Pain and Disability Index (SPADI) | at 3 weeks, 6 weeks, 3 months, 6 months, 9 months and 12 months
  It is a self-written questionnaire. It consists of twosubscales. The first assesses the importance of pain felt on five items. Pain scores range from 0 to 50. The second evaluates the difficulty of activities of daily living based on eight. Scores range from 0 to 80.questions

SECONDARY OUTCOMES:
pain using a visual analogue scale | at 3 weeks, 6 weeks, 3 months, 6 months, 9 months and 12 months
  It is a 100mm ruler that allows patients to rank their pain on a continuum from no pain to extreme pain. The patient places the indicator on a level that represents their current pain.
Active and passive range of motion | at 3 weeks, 6 weeks, 3 months, 6 months, 9 months and 12 months
  Active and passive range of motion is clinically assessed using a goniometer while standing. We measured abduction, extension and external rotation.

CONTACTS AND LOCATIONS:
Overall Officials: samia karkouri, professor, Study Chair — Mohammed V Souissi University
Locations (1):
- Faculty of medecine and pharmacy of rabat, Rabat, Morocco

IPD SHARING:
Plan to Share IPD: Yes
excell table of data
Supporting Information: Study Protocol, SAP
Time Frame: start january 2025 end may 2025
Access Criteria: doctors in the rehabilitation field can ask access by sending an email to the principal investigator